CLINICAL TRIAL: NCT04037501
Title: "Care Management for Caregivers of People With Dementia: Effectiveness of a Care Management System to Reduce Unmet Needs of Informal Caregivers of People With Dementia"
Brief Title: Effectiveness of a Care Management System to Reduce Unmet Needs of Informal Caregivers of People With Dementia
Acronym: GAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Collaborators: Gemeinsamer Bundesausschuss (GBA) (Unknown); University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Wolfgang Hoffmann, Site speaker, German Center for Neurodegenerative Diseases (DZNE)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GR009; 01VSF18030 (Other Grant/Funding Number: Gemeinsamer Bundesausschuss (GBA))
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Dementia; Caregiver Burnout; Carer Stress Syndrome; Relatives; Partner, Domestic
Keywords: Caregiver of people with dementia; Caregiver health; Care management system; Collaborative care; Informal care coordination; Dementia; Medical management; Unmet needs
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Care Management
- care as usual (No Intervention)

INTERVENTIONS:
Other: Care Management — A computerized Care Management System (CMS) will identify unmet needs of the informal caregiver of PwD and generates suggestions for interventions. Based on these, the treating physician develops an individualized treatment and care plan and assigns specific tasks to the care manager. Upon a home visit in the caregivers' home the care manager evaluates the need for additional tasks. Based on the complete list of tasks, the care manager initiates the implementation of respective actions. Via monthly telephone calls and optional home visits the care manager monitors the status of implementation and actively coordinates the support and care for the informal caregiver recommended intervention
  Arms: Intervention

SUMMARY:
The purpose of this study is to test the effectiveness of a computer assisted care management system to identify and reduce unmet needs for and to improve quality of life of informal caregivers of people with dementia.

DETAILED DESCRIPTION:
The identification of care needs of informal caregivers of people with dementia (PwD) at home is of particular importance to provide timely appropriate support and health care services to this vulnerable group. Family doctors and specialists have a key role in identifying the burden and care needs of informal caregivers. However, this often remains a challenge in everyday practice. In addition, the regionally available support and health care offers are often unknown. A computer-assisted care management system (CMS) can support the identification of unmet care needs and suggest individual, regional offers via a constantly updated database. On the basis of a standardized self-assessment, the VMS identifies personal, social, nursing and medical care needs of informal caregivers of PwD. The investigators apply the system in family and specialist practices as well as in memory clinics where it generates modularized recommendations for interventions based on predefined algorithms. The aim of the study is to test the effectiveness of a CMS to reduce the number of unmet care needs and to improve quality of life of informal caregivers of PwD. The study design is a cluster-randomized, controlled intervention study with two arms and two assessment times. The setting includes family and specialist practices for neurology and/ or psychiatry as well as memory clinics. The CMS will be used in the practices of the intervention group. Informal caregivers of PwD answer a self-administered questionnaire on a tablet PC. From the input, the system generates a list of unmet care needs based on predefined algorithms, and assigns these to individual intervention recommendations. The doctor evaluates each recommendation and forwards a validated list and possibly further intervention recommendations to a study assistant (Care Manager, CM). In a subsequent home visit, the care manager systematically collects additional information, specifies and concretizes the intervention recommendations and supports the informal caregivers of PwD in the implementation of the recommendations. In subsequent telephone contacts, the status of the implementation of the intervention recommendations will be discussed and the care manager coordinates the informal caregivers individual support. Patients of the control group will receive Care as Usual (CAU). After 6 months, a blinded, systematic, computer-based follow-up assessment will be conducted in both groups by hitherto uninvolved study assistants

ELIGIBILITY:
Inclusion Criteria:

* 18+ years
* main caregiver of a PwD (Hauptversorgungsperson)
* PwD lives at home
* written informed consent of caregiver

Exclusion Criteria:

* caregiver not living in the study region MV
* not able to provide written consent
* unable to fill out self-administered questionnaire an/or to be interviewed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in number of Unmet Needs | Baseline values assessed at time of visit to the physician (T0), Outcome value assessed 6 months later at concluding home visit (T6)
  A standardized assessment implemented as computer-assisted intervention management system (CMS) addresses caregiver burden, medical needs, home care needs, psychosocial needs (depression, sleep quality, pain, hearing, seeing, teeth problems, dementia related problems caused by PwD, medical aids). Based on predefined algorithms the CMS will generate a list of recommended intervention to address each of the unmet needs.
Change in Quality of Life | Baseline values assessed at time of visit to the physician (T0), Outcome value assessed 6 months later at concluding home visit (T6)]
  The questionnaire SF-12 (Short form of SF-36) will be used to assess quality of life. The SF-12 is a physical scale score that represents general health perception, physical functioning, physical role functioning, and pain. The mental health score represents emotional role functioning, mental well-being, negative affectivity, and social functioning. The mean score is set to 50. Scores higher than 50 indicate better physical or mental health than the mean while scores lower than 50 indicate worse physical mental health than the mean.

SECONDARY OUTCOMES:
Change in Caregiver Burden | Baseline values assessed at time of visit to the physician (T0), Outcome value assessed 6 months later at concluding home visit (T6)]
  Informal caregiver burden will be assessed using the 7-item (short) version of the Zarit-Burden Interview; ZBI-7. The short version ZBI is a caregiver self-report measure to examine burden which is associated with functional/behavioural impairments in the social, psychological and physiological context and home care situation.It contains 7 items using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly/Always). Total scores range from 0 indicating low burden to 88 indicating high burden.
Social Support | Baseline values assessed at time of visit to the physician (T0), Outcome value assessed 6 months later at concluding home visit (T6)
  Social support will be assessed using the Lubben Social Network Scale (LSNS). This scale is a self-report measure of social engagement including family and friends on a 12 item scale. Total scores ranging from 0 to 90. High scores indicate strong social networks.
Use of medical and non-medical services | : Baseline values assessed at time of visit to the physician (T0), Outcome value assessed 6 months later at concluding home visit (T6)]
  The use of medical and non-medical services will be assessed using the Questionnaire for the Use of Medical and Non-Medical Services in Old Age [Fragebogen zur Inanspruchnahme medizinischer und nicht-medizinischer Versorgungsleistungen im Alter". The FIMA examines socio-economic variables and other medical factors to determine health-related costs.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hoffmann, MD, Principal Investigator — German Center for Neurodegenerative Diseases (DZNE)
Locations (1):
- German Center for Neurodegenerative Diseases (DZNE), Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klein OA, Boekholt M, Afrin D, Dornquast C, Dreier-Wolfgramm A, Keller A, Michalowsky B, Zwingmann I, Teipel S, Thyrian JR, Kilimann I, Hoffmann W. Effectiveness of a digitally supported care management programme to reduce unmet needs of family caregivers of people with dementia: study protocol for a cluster randomised controlled trial (GAIN). Trials. 2021 Jun 16;22(1):401. doi: 10.1186/s13063-021-05290-w. PMID 34134744